CLINICAL TRIAL: NCT03601533
Title: Prospective Study of the Efficacy of Ultrasound-guided Genicular Nerve Block With Phenol for the Treatment of Chronic Pain Due to Knee Osteoarthritis
Brief Title: Ultrasound-guided Genicular Nerve Block With Phenol for the Treatment of Chronic Pain Due to Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, Professor, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Phenol
Record Dates: First submitted 2018-07-12; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Osteoarthritis, Knee; Chronic Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Phenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phenol (Other): Patients will undergo neurolysis of genicular nerves with 1,5 mL of 7% phenol in each of the genicular nerves (superior, medial and lateral).
  Interventions: Drug: Phenol

INTERVENTIONS:
Drug: Phenol — 1,5 mL of 7% phenol will be injected in each of genicular nerves (superior, medial and lateral).

SUMMARY:
Osteoarthritis (OA) is one of the most frequent causes of chronic pain, often intense, debilitating and responsible for a large percentage of the elderly. The disease affects about 10% of adults and the knees are the most affected joints. The diagnosis of OA in the knee is predominantly clinical, and can be confirmed by radiological examination. Systemic drugs are indicated before invasive procedures, but pharmacological therapies may offer limited benefits. Thermal radiofrequency lesions of genicular nerves has been used to relieve chronic knee pain, as adjuvant therapy, but with high costs and low availability in the public system. The use of phenol for peripheral analgesic blocks has emerged as a good option and at low cost and can be used in any service of Pain Treatment. The aim of the study is to evaluate the efficacy of 6% phenol for ultrasound-guided genicular nerves neurolysis for the treatment of patients with chronic knee pain due to osteoarthritis.

METHODS: A prospective study will be carried out with 15 patients with chronic pain (more than 4 months) and diagnosis of arthrosis by imaging, with pain intensity greater than 4 (from zero to 10) that will be submitted to ultrasound-guided genicular nerves block. The test block will be performed with 0.25% -1,5 mL bupivacaine on each nerve. Patients who present pain improvement> 50% will undergo neurolysis of genicular nerves with 1,5 mL of 7% phenol in each of the genicular nerves. After the procedure, the patients will be evaluated for 3 months in relation to the intensity of pain at rest and movement and duration of analgesia provided by the intervention, range of movements and functionality of the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the free, informed consent form
* Age over 18 years old
* Knee pain for more than six months without improvement with clinical treatment
* Clinical and imaging diagnosis (radiography) of knee osteoarthritis
* Moderate pain intensity (pain greater than 4, by the numerical scale).

Exclusion Criteria:

* Cognitive impairment or psychiatric disease
* Other causes of knee pain (trauma, complex regional pain syndrome)
* Puncture site infection
* Coagulopathy or use of anticoagulant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pain score | 15 days, 1 month, 2 months and 3 months after the procedure.
  Patients will be evaluated before the procedure (baseline) and for 3 months in relation to the intensity of pain at rest and movement . The numeric pain scale from 0 (best condition) to 10 (worst condition) will be used to evaluate the patients.

SECONDARY OUTCOMES:
Change from Baseline WOMAC score | 15 days, 1 month, 2 months and 3 months after the procedure
  Patients will be evaluated before the procedure (baseline) and for 3 months after the procedure in relation to the WOMAC score. The WOMAC range from 0 (best condition) to 100 ( worst condition).

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo HC Ferraro, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wong J, Bremer N, Weyker PD, Webb CA. Ultrasound-Guided Genicular Nerve Thermal Radiofrequency Ablation for Chronic Knee Pain. Case Rep Anesthesiol. 2016;2016:8292450. doi: 10.1155/2016/8292450. Epub 2016 Oct 16. PMID 27822391
- [Result] Bijlsma JW, Berenbaum F, Lafeber FP. Osteoarthritis: an update with relevance for clinical practice. Lancet. 2011 Jun 18;377(9783):2115-26. doi: 10.1016/S0140-6736(11)60243-2. PMID 21684382
- [Result] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Result] Brenner SS, Klotz U, Alscher DM, Mais A, Lauer G, Schweer H, Seyberth HW, Fritz P, Bierbach U. Osteoarthritis of the knee--clinical assessments and inflammatory markers. Osteoarthritis Cartilage. 2004 Jun;12(6):469-75. doi: 10.1016/j.joca.2004.02.011. PMID 15135143
- [Result] Yasar E, Kesikburun S, Kilic C, Guzelkucuk U, Yazar F, Tan AK. Accuracy of Ultrasound-Guided Genicular Nerve Block: A Cadaveric Study. Pain Physician. 2015 Sep-Oct;18(5):E899-904. PMID 26431143
- [Result] Gebhardt R, Wu K. Transversus abdominis plane neurolysis with phenol in abdominal wall cancer pain palliation. Pain Physician. 2013 May-Jun;16(3):E325-30. PMID 23703432
- [Result] Koyyalagunta D, Engle MP, Yu J, Feng L, Novy DM. The Effectiveness of Alcohol Versus Phenol Based Splanchnic Nerve Neurolysis for the Treatment of Intra-Abdominal Cancer Pain. Pain Physician. 2016 May;19(4):281-92. PMID 27228515
- [Result] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159